CLINICAL TRIAL: NCT05210829
Title: The Association Between Parent Anxiety and Sedation Anesthesia Doses in Pediatric Endoscopy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Elif Erdoğan Öngel, Elif Erdogan-Ongel, Saglik Bilimleri Universitesi
Other Study IDs: Sancaktepe Pediatric Endoscopy
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Anxiety; Anesthesia
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High Parent Anxiety: Stationary and Trait Anxiety Scale ≥ 44 points
  Interventions: Diagnostic Test: stationary and trait anxiety scale
- Low Parent Anxiety: Stationary and Trait Anxiety Scale < 44 points
  Interventions: Diagnostic Test: stationary and trait anxiety scale

INTERVENTIONS:
Diagnostic Test: stationary and trait anxiety scale — survey

SUMMARY:
Our study was planned as a prospective, single-center study between 20 January 2022 and 20 April 2022. All patients between the ages of 1-18 who will undergo upper or lower gastrointestinal endoscopy and their parents will be included in our study. All patients and parents whose family did not give consent to participate in the study will be excluded from the study. All patients will be seen by an anesthesiologist before the procedure and it will be stated that there is no harm in taking anesthesia. Anesthesia consent form will be given by the family. Study participation consent will be obtained from parents before starting the procedure. The patient's age, gender, height, weight, ASA score, the procedure to be performed, the parent's educational status, occupation and income level will be recorded. Children's anxiety will be evaluated with the "Modified Yale Preoperative Anxiety Scale (mYPAS)" in the presence of their parents 15-30 minutes before the procedure. The agitation that occurs when the patient leaves the families for processing, with the "Parental Separation Anxiety Scale"; Parental anxiety will be evaluated with the "Stationary and Trait Anxiety Scale" filled by families after the child is processed.

ELIGIBILITY:
Inclusion Criteria:

* All patients between the ages of 1-18 who will undergo upper or lower gastrointestinal endoscopy and their parents will be included in our study.

Exclusion Criteria:

* All patients and parents whose family did not give consent to participate in the study will be excluded from the study.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All patients between the ages of 1-18 who will undergo upper or lower gastrointestinal endoscopy and their parents.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-01-20 (Estimated); Primary Completion 2022-04-20 (Estimated); Study Completion 2022-04-20 (Estimated)

PRIMARY OUTCOMES:
Anesthesia agent dose | end of the gastrointestinal endoscopy

SECONDARY OUTCOMES:
Children's anxiety | before gastrointestinal endoscopy

IPD SHARING:
Plan to Share IPD: Undecided